CLINICAL TRIAL: NCT07131098
Title: Effectiveness of an Early Enteral Feeding Protocol on Clinical Outcomes in Critically Ill Patients: A Quasi-experimental Study
Brief Title: Early Enteral Feeding and Clinical Outcomes in ICU Patients
Acronym: EEFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loai Muawiah Zabin (Other)
Responsible Party: Sponsor-Investigator, Loai Muawiah Zabin, Faculty Member, Arab American University, Arab American University (Palestine)
Organization: Arab American University (Palestine) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAUP-EEFP-ICU-2024
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Enteral Nutrition; Intensive Care Unit ICU; Nutritional Support; Feeding Protocol
Keywords: Early enteral feeding; ICU nutrition; Critically ill patients; Quasi-experimental study; Palestine; Protocol-based nutrition; Clinical outcomes; Nutritional therapy; Mechanical ventilation; Length of ICU stay; Glasgow Coma Scale (GCS); Laboratory outcomes; Bicarbonate; Sodium; Platelets; Hemoglobin
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either an experimental group, receiving early enteral feeding per a structured protocol, or a control group, receiving standard nutritional care. Grouping was based on period of admission to minimize selection bias.
Masking Description: This was an open-label study. Neither the care providers nor the participants were blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Enteral Feeding Protocol (Experimental): Participants in this group received early enteral nutrition initiated within 24-48 hours of ICU admission, based on a structured feeding protocol. The protocol followed international guidelines (ASPEN/ESPEN) and was implemented by ICU staff with training and monitoring support.
  Interventions: Other: Early Enteral Feeding Protocol
- Standard Nutritional Care (Other): Participants in this group received standard ICU nutritional care without the implementation of the early enteral feeding protocol. Feeding initiation and type were left to physician discretion based on clinical judgment and routine hospital practices.
  Interventions: Other: Standard Nutritional Care

INTERVENTIONS:
Other: Early Enteral Feeding Protocol — Early enteral nutrition was initiated within 24-48 hours of ICU admission based on a structured protocol aligned with ASPEN and ESPEN guidelines. The protocol defined target caloric goals, methods of tube feeding initiation, rate advancement, and monitoring procedures. Nurses and ICU staff were trained in protocol implementation. The goal was to optimize nutrition early in critical illness to improve clinical outcomes such as ICU length of stay, ventilator dependence, and physiological stability.
  Arms: Early Enteral Feeding Protocol
Other: Standard Nutritional Care — Patients in the control group received standard nutritional care per routine hospital practices. Initiation and progression of feeding were left to the discretion of the attending physician and nursing staff, without the use of a structured protocol or defined early feeding timeline.
  Arms: Standard Nutritional Care

SUMMARY:
This study evaluated the effectiveness of an early enteral feeding protocol in critically ill adult patients admitted to an Intensive Care Unit (ICU). The intervention involved initiating enteral nutrition within 24-48 hours of ICU admission. Clinical outcomes such as ICU length of stay, ventilator dependency, and selected laboratory values were compared between patients who received early enteral feeding and those who received standard nutritional care. The study was conducted at Jenin Governmental Hospital in Palestine between January and April 2024, with 80 adult participants.

DETAILED DESCRIPTION:
This is a retrospectively registered, quasi-experimental study that investigated the clinical impact of implementing an early enteral feeding protocol in a critical care setting. Conducted in Jenin Governmental Hospital, Palestine, the research explored how protocolized early nutritional support affects physiological recovery and ICU-related outcomes in critically ill adult patients.

The study was motivated by the well-established role of early enteral nutrition in maintaining gut integrity, supporting immune function, and reducing complications in ICU patients. Despite international guidelines recommending its use within 24-48 hours of ICU admission, early enteral feeding remains underutilized in many low-resource healthcare settings. Factors contributing to this gap include variability in clinical practice, limited institutional protocols, and staff training constraints.

This investigation was carried out between January and April 2024 and followed rigorous ethical standards, with Institutional Review Board approval from Arab American University (Reference: R-2024/B/85/N). Patients were grouped based on the time period of admission into either a protocol-based early feeding group or a standard care group. Intervention fidelity was maintained through a pre-defined feeding protocol implemented by ICU staff after appropriate orientation and monitoring.

The study contributes to the growing body of evidence supporting structured nutritional protocols in ICUs and highlights the feasibility and benefits of such interventions in middle-income and resource-constrained settings. The data gathered and analyzed provide a foundation for future policy development aimed at standardizing nutritional support for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Admitted to the ICU and eligible for enteral feeding
* Expected to stay in the ICU for more than 48 hours
* Able to initiate enteral feeding within 24-48 hours of ICU admission
* Informed consent obtained from the patient or legal guardian

Exclusion Criteria:

* Pregnant or lactating women
* Patients with gastrointestinal bleeding or obstruction
* Patients undergoing gastrointestinal surgery or with short bowel syndrome
* Diagnosed with COVID-19 during admission
* End-of-life care patients or those with do-not-resuscitate (DNR) orders
* Refusal to participate or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Length of ICU Stay (in days) | Through ICU discharge, up to 7 days
  Duration of patient stay in the intensive care unit, measured in full days from admission to discharge.

SECONDARY OUTCOMES:
Glasgow Coma Scale (GCS) Score | Daily for up to 7 days.
  Assessment of neurological status using the GCS; higher scores indicate better consciousness levels.
Hemoglobin Level (g/dL) | Day 1 and Day 7 of ICU stay
  Laboratory measure of hemoglobin concentration as an indicator of oxygen-carrying capacity and blood loss.
Bicarbonate (HCO₃) Level (mEq/L) | Day 1 and Day 7 of ICU stay
  Blood bicarbonate levels used to assess acid-base balance in critically ill patients.
Platelet Count (×10³/μL) | Day 1 and Day 7 of ICU stay
  Platelet concentration is measured from a complete blood count to evaluate clotting potential and bone marrow function.
Calcium Level (mg/dL) | Day 1 and Day 7 of ICU stay
  Measurement of serum calcium levels to assess electrolyte balance and nutritional status.
Mechanical Ventilation Duration (in days) | Through ICU discharge, up to 7 days
  Total number of days the patient required mechanical ventilation during ICU stay.
Fraction of Inspired Oxygen (FiO₂) Requirement (%) | Daily for up to 7 days
  Daily measurement of the fraction of inspired oxygen (%) required by patients during mechanical ventilation in the ICU, used to assess respiratory support needs. Values will be recorded once daily and analyzed as mean values over the ICU stay.
Positive End-Expiratory Pressure (PEEP) Requirement (cmH₂O) | Daily for up to 7 days
  Daily measurement of positive end-expiratory pressure (PEEP, in cmH₂O) applied during mechanical ventilation in the ICU, used to assess respiratory support needs. Values will be recorded once daily and analyzed as mean values over the ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Mahameed, Master, Principal Investigator — Arab American University (Palestine); Sajed Ghawadra, PhD, Study Chair — Arab American University (Palestine)
Locations (1):
- Jenin Governmental Hospital, Jenin, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during this study will not be shared publicly due to ethical and legal restrictions. The study involved critically ill patients in an intensive care setting, and data sharing was not included in the original informed consent or ethics approval. Ensuring patient confidentiality and privacy remains a top priority.